CLINICAL TRIAL: NCT04898101
Title: Absolute Bioavailability, Pharmacokinetics, Excretion, and Metabolism of [14C]Acp-196 (Acalabrutinib) in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of [14C]Acp-196 (Acalabrutinib) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-009
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: ACP-196; Acalabrutinib; [14C]Acp-196; Healthy participants; Volunteers; Adults; Pharmacokinetics; PK; Bioavailability; Excretion; Metabolism
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive a single 100 mg oral capsule dose of acalabrutinib and at 58 minutes postdose, participants will receive a single microtracer (<10 μg; <=1 μCi) [14C]ACP-196 as a 5 mL IV push over 2 minutes.
  Interventions: Drug: Acalabrutinib; Drug: Microtracer [14C]ACP-196
- Cohort 2 (Experimental): Participants will receive a single 100 mL oral solution of acalabrutinib, 1 mg/mL oral solution containing a microtracer dose (<10 μg; <=1 μCi) of [14C]ACP-196.
  Interventions: Drug: Microtracer [14C]ACP-196

INTERVENTIONS:
Drug: Acalabrutinib — Participants in Cohort 1 will receive a single 100 mg oral capsule dose of acalabrutinib on Day 1.
  Other Names: ACP-196
  Arms: Cohort 1
Drug: Microtracer [14C]ACP-196 — Participants in Cohort 1 will receive a single microtracer (<10 μg; ≤1 μCi) IV solution dose of [14C]ACP-196 as a 5-mL IV push over 2 minutes on Day 1. Participants in Cohort 2 will receive a single 100 mL dose of acalabrutinib 1 mg/mL oral solution containing a microtracer dose (<10 μg; ≤1 μCi) of [14C]ACP-196 on Day 1.

SUMMARY:
This study is to determine the absolute bioavailability of oral acalabrutinib and intravenous (IV) PK of [14C]ACP-196.

DETAILED DESCRIPTION:
This is 2-cohort study. Screening period will be within 28 days before the dose. In the treatment period, participants in Cohort 1 will receive a single 100 mg oral capsule dose of acalabrutinib and at 58 minutes postdose of acalabrutinib will receive a single microtracer (<10 μg; <=1 μCi) [14C]ACP-196 as a 5 mL IV push over 2 minutes; and participants in Cohort 2 will receive a single 100 mL oral solution of acalabrutinib (1 mg/mL oral solution containing a microtracer dose (<10 μg; <=1 μCi) of [14C]ACP-196). Cohort 1 participants will be confined continuously from Check-in until Day 5 and Cohort 2 participants will be confined continuously from Check-in until Day 8.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine-containing products within 3 months before Check-in and during the entire study
* Body mass index (BMI) >= 18.5 to <= 29.9 kg/m^2 at Screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the investigator
* Women must be of non-childbearing status and have negative serum pregnancy test results at Screening and Check-in
* Male participants must be willing to use protocol specified contraception methods
* A minimum of 1 bowel movement per day (Cohort 2 only)

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History of any illness that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* Presence of any clinically significant, ongoing systemic bacterial, fungal, or viral infections in the opinion of the investigator
* History or presence of alcoholism or drug abuse within the past 2 years before Screening
* History of bleeding diathesis
* Any clinically significant condition that may affect acalabrutinib absorption in the opinion of the investigator, including gastric restrictions and bariatric surgery (eg, gastric bypass)
* History or presence of clinically significant thyroid disease, in the opinion of the investigator
* Women who are pregnant, breastfeeding, or lactating
* Positive test for selected drugs of abuse at Screening and at Check-in
* Known history of human immunodeficiency virus (HIV), serologic status reflecting active or past history of hepatitis B or C infection, or any uncontrolled active systemic infection
* Supine blood pressure is < 90/40 mmHg or > 140/90 mmHg at Screening
* Supine pulse is < 40 beats per minute or > 99 beats per minute at Screening
* Have been on a diet incompatible with the on-study diet, in the opinion of the Investigator, within the 28 days before the dose of study drug, and throughout the study
* Unable to refrain from or anticipates the use of any drugs, including prescription and non-prescription medications
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months before Check-in
* Exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal) or current employment in a job requiring radiation exposure monitoring, with either being within 12 months before Check-in
* Poor peripheral venous access
* Unwilling to consume trace amounts of ethanol (alcohol) that may be present in the dose formulation
* History or presence of liver disease or cholecystectomy and Clostridium difficile associated diarrhea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) of Acalabrutinib for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
Area Under the Concentration-time Curve From Hour 0 to the Last Quantifiable Concentration (AUC0-t) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Area Under the Concentration-time Curve From Hour 0 to Hour 12 (AUC0-12h) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Area Under the Concentration-time Curve From Hour 0 to Hour 72 (AUC0-72h) of Acalabrutinib and [14C]ACP-196 for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
Area Under the Concentration-time Curve From Hour 0 to Hour 168 (AUC0-168h) of Acalabrutinib and [14C]ACP-196 for Cohort 2 | Cohort 2: 0, 15, 30, 45, 60, 75, 90 min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hrs postdose
Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Percent of AUC0-inf Extrapolated (AUC%extrap) of ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Maximum Observed Concentration (Cmax) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Time to Maximum Observed Concentration (tmax) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Apparent Terminal Elimination Half-life (t1/2) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Apparent Terminal Elimination Rate Constant (λz) of Acalabrutinib and [14C]ACP-196 for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Apparent Total Plasma Clearance (CL/F) of Acalabrutinib for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Total Plasma Clearance (CL) of [14C]ACP-196 for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Acalabrutinib for Cohort 1 and Cohort 2 | Cohort 1: 0, 15, 30, 45, 58min; post IV at 0, 5, 10, 15, 20, 30min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96hrs; Cohort 2: 0, 15, 30, 45, 60, 75, 90min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168hrs postdose
Volume of Distribution During the Terminal Phase (Vz) of [14C]ACP-196 for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
Volume of Distribution at Steady State (Vss) of [14C]ACP-196 for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
Mean Residence Time (MRT) of [14C]ACP-196 for Cohort 1 | Cohort 1: 0, 15, 30, 45, 58 min; post IV at 0, 5, 10, 15, 20, 30 min; and post oral dose at 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96 hrs
ACP-196:total 14C AUC0-inf Ratio for Cohort 2 | Cohort 2: 0, 15, 30, 45, 60, 75, 90 min, and at 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hrs postdose
Ratio of Whole Blood to Plasma AUC0-∞ for Total Radioactivity for Cohort 2 | Urine: -12 to 0 (before dose within 20 minutes), 0 to 6 hrs, 6 to 12 hrs, 12 to 24 hrs, and 24-hr intervals through 168 hrs postdose; Feces: predose (within 24 hours of dosing), 0 to 24 hrs postdose, and 24-hr intervals through 168 hrs postdose
Cumulative Amount of Drug Excreted in Urine (Aeu) of Acalabrutinib and [14C]ACP-196 for Cohort 1 | Urine at -12 to 0 (before dose, up to the last void within 20 minutes before oral dosing), 0 to 6 hrs, 6 to 12 hrs, 12 to 24hrs, 24 to 48hrs, and 48 to 72hrs post oral dose
Renal Clearance (CLR) of Acalabrutinib and [14C]ACP-196 for Cohort 1 | Urine at -12 to 0 (before dose, up to the last void within 20 minutes before oral dosing), 0 to 6 hrs, 6 to 12 hrs, 12 to 24hrs, 24 to 48hrs, and 48 to 72hrs post oral dose
Cumulative Percent of Dose Excreted in Urine (%feu) of Acalabrutinib and [14C]ACP-196 for Cohort 1 | Urine at -12 to 0 (before dose, up to the last void within 20 minutes before oral dosing), 0 to 6 hrs, 6 to 12 hrs, 12 to 24hrs, 24 to 48hrs, and 48 to 72hrs post oral dose
Cumulative Amount of Drug Excreted in Urine of Acalabrutinib and Urine and Fecal (Ae) of [14C]ACP-196 for Cohort 2 | Urine: -12 to 0 (before dose within 20 minutes), 0 to 6 hrs, 6 to 12 hrs, 12 to 24 hrs, and 24-hr intervals through 168 hrs postdose; Feces: predose (within 24 hours of dosing), 0 to 24 hrs postdose, and 24-hr intervals through 168 hrs postdose
Cumulative Percent of Dose Excreted in Urine of Acalabrutinib and Urine and Fecal (%fe) of [14C]ACP-196 for Cohort 2 | Urine: -12 to 0 (before dose within 20 minutes), 0 to 6 hrs, 6 to 12 hrs, 12 to 24 hrs, and 24-hr intervals through 168 hrs postdose; Feces: predose (within 24 hours of dosing), 0 to 24 hrs postdose, and 24-hr intervals through 168 hrs postdose

SECONDARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Cohort 1: From Day 1 through Day 5; Cohort 2: From Day 1 through Day 8
Incidence of Abnormal Clinical Laboratory Parameters Reported as TEAEs | Cohort 1: From Day 1 through Day 5; Cohort 2: From Day 1 through Day 8
Incidence of Abnormal Vital Signs and Physical Examinations Reported as TEAEs | Cohort 1: From Day 1 through Day 5; Cohort 2: From Day 1 through Day 8
Incidence of Abnormal ECGs Reported as TEAEs | Cohort 1: From Day 1 through Day 5; Cohort 2: From Day 1 through Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Priti Patel, Study Director — Acerta Pharma BV
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home